CLINICAL TRIAL: NCT05754112
Title: Dissecting the Role of B Lymphocytes in the Loss of Immunological Tolerance and Disease Resolution Through JAK Signaling In Rheumatoid Arthritis
Brief Title: JAK-i on RA B-lymphocytes Tolerance and Disease Resolution Through JAK Signaling In Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Gremese Elisa, Prof., Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4109
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- ACPA/RFpos asyntomatic individuals: ACPA and/or RF positive individuals without active arthritis
  Interventions: Other: B lymphocyte profiling
- Naive Active RA: Treatment-naive active RA (disease duration<1 year)
  Interventions: Other: B lymphocyte profiling
- Resistant RA: Active despite treatment RA
  Interventions: Other: B lymphocyte profiling
- Remission RA: RA in sustained clinical and ultrasound remission
  Interventions: Other: B lymphocyte profiling
- Control Group: Individuals asymptomatic for joint inflammation without ACPA/RF positivity
  Interventions: Other: B lymphocyte profiling

INTERVENTIONS:
Other: B lymphocyte profiling — All individuals will undergo peripheral venous blood sampling and ultrasound-guided synovial tissue biopsy following a standardized procedure. B-lymphocytes will be sorted from PBMCs isolated by Ficoll gradient method using magnetic CD19-microbeads whereas tissue B-lymphocytes will be isolated from synovial tissue biopsies digested with Liberase. CD19 positive cells from PBMC will be incubated with pro-inflammatory molecules in presence or absence of Ubadacitinib. After stimulation, CD19 positive cells will be collected and processed for single cell RNA sequencing. Moreover, the impact of JAK-1 selective inhibition on B-lymphocyte cultures stimulation will be tested using ELISA method for the assessment of cytokines/chemokines production. Synovial tissue and synovial tissue B-lymphocyte subpopulations will be assessed through FACS analysis using IgD/CD27 classification. Finally, we will compare the transcriptomic profile of synovial tissue B lymphocytes from 5 subject groups.

SUMMARY:
The study will reveal the transcriptomic signature linked to the aberrant activation of B lymphocytes in RA identifying novel molecular potential targets for inflammation resolution and immune tolerance promotion. The combination with B lymphocytes phenotyping will dissect the impact of the identified genes on B lymphocyte maturation and activation in RA. Moreover, in vitro study on B lymphocyte cultures using selective JAK1 inhibition will reveal, at deeper level, its transcriptomic effect on RA B lymphocytes activation profile and phenotype, providing the discovery of new biomarkers of the loss of immunological tolerance, active disease and long lasting disease remission.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent. Before any study procedures are performed,subjects will have the details of the study described to them, and they will be given a written informed consent document to read. Then, if subjects consent to participate in the study, they will indicate that consent by signing and dating the informed consent document in the presence of trained study personnel.
2. Patients fulfilling classification criteria for Rheumatoid Arthritis (2010 ACR/EULARclassification criteria)
3. Age: 18-70 years
4. For preclinical cohort: Individuals with positivity for ACPA or IgM/IgA RF without clinical signs of arthritis, whose positivity is not related to other concomitant pathologic conditions.
5. For naive to treatment cohort: RA patients without previous exposure to conventional DMARDs or biologic/targeted synthetic-DMARDs.
6. For resistant to treatment cohort: RA patients with failure to previous conventionalDMARDs for inadequate response or side effects.
7. For remission RA cohort: RA patients in sustained clinical and ultrasound remission as stated in section 3.3.1.
8. For healthy control cohort: Healthy donors will be aged from 18 to 70 years.

Exclusion Criteria:

1. Severe and uncontrolled infections such as sepsis and opportunistic infections.
2. Patients who are currently included in any interventional clinical trial in RA.
3. RA patients in therapy with other biologics.
4. Healthy donors receiving anti-inflammatory drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is an interventional research without experimental drug which will be performed at the Division of Clinical Immunology of the Fondazione Policlinico Universitario A. Gemelli IRCCS in Rome, Italy, where patients with Rheumatoid Arthritis will undergo to synovial tissue inflammation assessment through minimally invasive US-guided synovial tissue biopsy.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-29 (Actual); Primary Completion 2023-05-02 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Peripheral blood and synovial tissue B lymphocyte atlas | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Immunology, Fondazione Policlinico Universitario A. Gemelli-IRCCS, Rome, Italy